CLINICAL TRIAL: NCT00515554
Title: HD18 for Advanced Stages in Hodgkins Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Engert, Prof., University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HD18
Record Dates: First submitted 2007-08-10; First posted 2007-08-13 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Hodgkins Lymphoma
Keywords: Hodgkin lymphoma; PET; advances stages; Rituximab
MeSH Terms: conditions — Hodgkin Disease | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Active Comparator): 8 cycles BEACOPPesc
  Interventions: Drug: BEACOPP escalated
- B (Experimental): 8 cycles BEACOPPesc plus rituximab
  Interventions: Drug: Rituximab; Drug: BEACOPP escalated
- C (Active Comparator): 8 cycles BEACOPPesc
  Interventions: Drug: BEACOPP escalated
- D (Experimental): 4 cycles BEACOPPesc
  Interventions: Drug: BEACOPP escalated

INTERVENTIONS:
Drug: Rituximab — addition of Rituximab to BEACOPP escalated
  Arms: B
Drug: BEACOPP escalated — chemotherapy with BEACOPP escalated

SUMMARY:
This study is designed to test:

1. in patients with negative positron-emission tomography (PET) after 2 cycles of BEACOPPesc chemotherapy: whether the number of cycles can be reduced without compromising progression free survival (PFS) (2 further cycles vs. 6 further cycles)
2. for patients with positive PET after 2 cycles: whether intensifying BEACOPPesc chemotherapy by adding Rituximab improves PFS.

ELIGIBILITY:
Inclusion Criteria:

* Hodgkin Lymphoma (histologically proven)
* CS (PS) IIB with one or both of the risk factors:

  * bulky mediastinal mass (> 1/3 of maximum transverse thorax diameter)
  * extranodal involvement
* CS (PS) III, IV
* Written informed consent

Exclusion Criteria:

* Leucocytes < 3000/µl
* Platelets < 100000/µl
* Hodgkin´s lymphoma as "composite lymphoma"
* Activity index (WHO) < grade 2

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1500 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 5 years

SECONDARY OUTCOMES:
Overall Survival | 5 years
acute toxicity | 5 years
late toxicity | 5 years
CR-rate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, Prof., Principal Investigator — University of Cologne
Locations (1):
- 1st Dept. of Medicine, Cologne University Hospital, Cologne, Germany

REFERENCES:
- [Derived] Lommen M, Weindler JJ, Jablonski J, Rosenbrock J, Borchmann P, Behringer K, Roth KS, Ufton D, Dietlein M, Kobe C, Ferdinandus J. Association between metabolic tumor burden and health-related quality of life in patients with classic Hodgkin lymphoma. Eur J Nucl Med Mol Imaging. 2025 Oct 11. doi: 10.1007/s00259-025-07569-5. Online ahead of print. PMID 41074963
- [Derived] Kreuzberger N, Goldkuhle M, von Tresckow B, Kobe C, Sickinger MT, Monsef I, Skoetz N. Positron emission tomography-adapted therapy for first-line treatment in adults with Hodgkin lymphoma. Cochrane Database Syst Rev. 2025 Mar 26;3(3):CD010533. doi: 10.1002/14651858.CD010533.pub3. PMID 40135712
- [Derived] Kreissl S, Goergen H, Buehnen I, Kobe C, Moccia A, Greil R, Eichenauer DA, Zijlstra JM, Markova J, Meissner J, Feuring-Buske M, Soekler M, Beck HJ, Willenbacher W, Ludwig WD, Pabst T, Topp MS, Hitz F, Bentz M, Keller UB, Kuhnhardt D, Ostermann H, Hertenstein B, Aulitzky W, Maschmeyer G, Vieler T, Eich H, Baues C, Stein H, Fuchs M, Diehl V, Dietlein M, Engert A, Borchmann P; German Hodgkin Study Group. PET-guided eBEACOPP treatment of advanced-stage Hodgkin lymphoma (HD18): follow-up analysis of an international, open-label, randomised, phase 3 trial. Lancet Haematol. 2021 Jun;8(6):e398-e409. doi: 10.1016/S2352-3026(21)00101-0. PMID 34048679
- [Derived] Kobe C, Goergen H, Baues C, Kuhnert G, Voltin CA, Zijlstra J, Hoekstra O, Mettler J, Drzezga A, Engert A, Borchmann P, Dietlein M. Outcome-based interpretation of early interim PET in advanced-stage Hodgkin lymphoma. Blood. 2018 Nov 22;132(21):2273-2279. doi: 10.1182/blood-2018-05-852129. Epub 2018 Aug 30. PMID 30166329
- [Derived] Voltin CA, Goergen H, Baues C, Fuchs M, Mettler J, Kreissl S, Oertl J, Klaeser B, Moccia A, Drzezga A, Engert A, Borchmann P, Dietlein M, Kobe C. Value of bone marrow biopsy in Hodgkin lymphoma patients staged by FDG PET: results from the German Hodgkin Study Group trials HD16, HD17, and HD18. Ann Oncol. 2018 Sep 1;29(9):1926-1931. doi: 10.1093/annonc/mdy250. PMID 30010775
- [Derived] Borchmann P, Goergen H, Kobe C, Lohri A, Greil R, Eichenauer DA, Zijlstra JM, Markova J, Meissner J, Feuring-Buske M, Huttmann A, Dierlamm J, Soekler M, Beck HJ, Willenbacher W, Ludwig WD, Pabst T, Topp MS, Hitz F, Bentz M, Keller UB, Kuhnhardt D, Ostermann H, Schmitz N, Hertenstein B, Aulitzky W, Maschmeyer G, Vieler T, Eich H, Baues C, Stein H, Fuchs M, Kuhnert G, Diehl V, Dietlein M, Engert A. PET-guided treatment in patients with advanced-stage Hodgkin's lymphoma (HD18): final results of an open-label, international, randomised phase 3 trial by the German Hodgkin Study Group. Lancet. 2017 Dec 23;390(10114):2790-2802. doi: 10.1016/S0140-6736(17)32134-7. Epub 2017 Oct 20. PMID 29061295
- [Derived] Borchmann P, Haverkamp H, Lohri A, Mey U, Kreissl S, Greil R, Markova J, Feuring-Buske M, Meissner J, Duhrsen U, Ostermann H, Keller U, Maschmeyer G, Kuhnert G, Dietlein M, Kobe C, Eich H, Baues C, Stein H, Fuchs M, Diehl V, Engert A. Progression-free survival of early interim PET-positive patients with advanced stage Hodgkin's lymphoma treated with BEACOPPescalated alone or in combination with rituximab (HD18): an open-label, international, randomised phase 3 study by the German Hodgkin Study Group. Lancet Oncol. 2017 Apr;18(4):454-463. doi: 10.1016/S1470-2045(17)30103-1. Epub 2017 Feb 22. PMID 28236583
- [Derived] Sauer M, Plutschow A, Jachimowicz RD, Kleefisch D, Reiners KS, Ponader S, Engert A, von Strandmann EP. Baseline serum TARC levels predict therapy outcome in patients with Hodgkin lymphoma. Am J Hematol. 2013 Feb;88(2):113-5. doi: 10.1002/ajh.23361. Epub 2012 Dec 8. PMID 23225085